CLINICAL TRIAL: NCT04963556
Title: Effects of Red Bull® on the Effects of Moderate Endurance Training Measured by Haemodynamic Parameters
Brief Title: Effects of Red Bull® on the Effects of Training and Haemodynamic Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Arno Schmidt-Trucksäss, Prof. Dr. med., University of Basel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017-01079
Record Dates: First submitted 2020-11-13; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Effects of; Food, Allergic

STUDY DESIGN:
Who Masked: Participant
Masking Description: Blinded to verum or placebo drink
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red Bull (Experimental): Drinking of 355 ml Red Bull
  Interventions: Dietary Supplement: Red Bull
- Placebo (Placebo Comparator): Drinking of 355 ml sweetened water
  Interventions: Dietary Supplement: Red Bull

INTERVENTIONS:
Dietary Supplement: Red Bull — Drinking of Red Bull before exercise
  Other Names: Placebo

SUMMARY:
Background:

The consumption of Energy Drinks (EDs) can acutely lead to negative side effects, such as raised blood pressure and impaired endothelial function. Nevertheless, they are sold worldwide and are often consumed before physical activity (PA). In contrast to the blood pressure elevating effect of EDs, PA leads to a reduction of blood pressure. The effect of ED consumption on blood pressure response during and after endurance training is currently unresolved.

Methods:

A total of 23 participants (eleven men, twelve women) were evaluated in the intervention study with a blinded Cross-Over Design. They consumed on two different days either 355 ml Red Bull (RB) or 355 ml Placebo (Pla) in randomised order. The peripheral (PBP) and central blood pressure (CBP) were measured before, during and after a 30-minute aerobic endurance training, by the Schiller BR-102 plus PWA device.

DETAILED DESCRIPTION:
Background:

The consumption of Energy Drinks (EDs) can acutely lead to negative side effects, such as raised blood pressure and impaired endothelial function. Nevertheless, they are sold worldwide and are often consumed before physical activity (PA). In contrast to the blood pressure elevating effect of EDs, PA leads to a reduction of blood pressure. The effect of ED consumption on blood pressure response during and after endurance training is currently unresolved.

Methods:

A total of 23 participants (eleven men, twelve women) were evaluated in the intervention study with a blinded Cross-Over Design. They consumed on two different days either 355 ml Red Bull (RB) or 355 ml Placebo (Pla) in randomised order. The peripheral (PBP) and central blood pressure (CBP) were measured before, during and after a 30-minute aerobic endurance training, by the Schiller BR-102 plus PWA device.

ELIGIBILITY:
Inclusion Criteria:

* No known cardiovascular diseases such as arterial hypertension and diabetes mellitus.
* No ophthalmological diseases such as glaucoma or macular degeneration.
* No regular medication
* No vasodilator abuse for 24 h before the respective intervention (e.g. smoking, use of stimulants, β-blockers).
* No pregnancy (anamnestic)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2017-06-18 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Effect on blood pressure | 24 hours
  Effect on systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Pulse wave velocity | 24 hours
  central pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Arno Schmidt-Trucksäss, MD, Principal Investigator — University of Basel
Locations (1):
- University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No